CLINICAL TRIAL: NCT04202055
Title: Immunologic Biomarker Profile of Cerebrospinal Fluid
Acronym: BIOMOG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2017-01/ET-01
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Neuromyelitis optica with anti-MOG
  Interventions: Other: Biomarker analysis
- Patients with Neuromyelitis optica with anti-AQP4
  Interventions: Other: Biomarker analysis
- Seronegative patients with Neuromyelitis optica
  Interventions: Other: Biomarker analysis
- Patients with recurrent-remitting multiple sclerosis: Patients with recurrent-remitting multiple sclerosis with medullary or optic involvement
  Interventions: Other: Biomarker analysis
- Progressive multiple sclerosis patients
  Interventions: Other: Biomarker analysis
- Symptomatic controls
  Interventions: Other: Biomarker analysis

INTERVENTIONS:
Other: Biomarker analysis — Detection of biomarker in cerebrospinal fluid

SUMMARY:
The aim of this study was the describe the Immunologic biomarker profile of cerebrospinal fluid in multiple sclerosis patients

ELIGIBILITY:
Inclusion Criteria:

* patients who have had neuromyelitis ptica with anti-AQP4 antibodies, or anti- Myelin Oligodendrocyte Glycoprotein antibodies, or double seronegative antibodies.
* Neuromyelitis Optica patients have been prospectively included in the OFSEP collection
* Multiple sclerosis patients, isolated myelitis or optic neuritis patients, and symptomatic controls whose samples will come from the "NEURO" collection of the Hospital Biological Collections Center,
* Patients have given their free consent for use of their samples in research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples stored from the NOMADMUS cohort in the OFSEP collection and the NEURO collection from the Centre de Collections Biologiques Hospitalières
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Level of glial fibrillar acidic protein in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of chitinase-3-like protein 1 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of neurofilament in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin-6 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin-8 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of C-X-C motif ligand (CXCL-13) in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of Matrix metalloproteinase-9 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of Soluble CD27 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin 10 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin 17A in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin 1B in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of monocyte chemoattractant protein-1 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of soluble intercellular adhesion molecule-1 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay
Level of soluble vascular cell adhesion molecule-1 in cerebrospinal fluid in patients with Neuromyelitis Optica with anti- Myelin Oligodendrocyte Glycoprotein | Baseline
  enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
Level of glial fibrillar acidic protein in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of chitinase-3-like protein 1 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of neurofilament in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin-6 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin-8 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of C-X-C motif ligand (CXCL-13) in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of Matrix metalloproteinase-9 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of Soluble CD27 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin 10 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin 17A in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of Interleukin 1B in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of monocyte chemoattractant protein-1 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of soluble intercellular adhesion molecule-1 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay
Level of soluble vascular cell adhesion molecule-1 in cerebrospinal fluid in each group | Baseline
  enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France